CLINICAL TRIAL: NCT04251988
Title: The Effectiveness of Virtual Reality (VR) to Reduce Pain and Anxiety During Genitourinary (GU) Scans
Brief Title: VR to Reduce Pain and Anxiety During GU Scans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Andy Y. Chang, Attending Physician; Vice Chief, Division of Pediatric Urology, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHLA-19-00403
Record Dates: First submitted 2020-01-23; First posted 2020-02-05 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Urologic Diseases; Urogenital Disease; Vesico-Ureteral Reflux
Keywords: virtual reality, voiding cystourethrogram, catheterization
MeSH Terms: conditions — Urologic Diseases; Urogenital Diseases; Vesico-Ureteral Reflux

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard of Care (No VR) Randomization (No Intervention): Patients will receive standard of care during catheterization, which includes caregiver presence in the room and Child Life Specialists in the room, if desired, and does not include virtual reality.
- VR Randomization (Experimental): Patients will receive virtual reality in addition to standard of care.
  Interventions: Device: Oculus Go VR

INTERVENTIONS:
Device: Oculus Go VR — virtual reality headset
  Arms: VR Randomization

SUMMARY:
This study aims to test the effectiveness of virtual reality (VR) in reducing pain and anxiety in children undergoing voiding cystourethrograms (VCUG) at Children's Hospital Los Angeles (CHLA). A voiding cystourethrogram is a genitourinary diagnostic scan that provides important urological information, specifically the filling and releasing of the bladder. This information can help diagnose urological issues in children. However, this procedure requires catheterization, which is understood to be a painful and anxiety-provoking procedure. This study will test the effectiveness of VR as a non-pharmaceutical intervention to relieve pain and anxiety in pediatric patients undergoing VCUGs.

DETAILED DESCRIPTION:
Background: VCUGs are genitourinary diagnostic scans that provide valuable medical information for pediatric patients with urological issues. However, these scans require catheterization, which can be anxiety-provoking, painful, and in some cases traumatic. Previous studies have assessed the use of pharmacological agents to address pain and anxiety during these procedures, but few studies exist examining non-pharmacological interventions in a methodologically rigorous way. As pharmacological interventions are associated with numerous side effects, and may not be appropriate for all pediatric patients, effective non-pharmacological interventions are needed for patients undergoing VCUGs.

Aims: This study aims to determine the effectiveness of virtual reality (VR) in reducing pain and anxiety among children undergoing VCUGs at CHLA. This study will also assess patient, parent, and provider satisfaction with VR, and ease of completing VCUGs using VR vs. the standard of care.

Study Population: CHLA patients aged 5-21 years receiving VCUGs at CHLA. Methods: A stratified randomization scheme will be used to assign patients aged 5-21 undergoing VCUG scans to receive the standard of care (i.e. caregiver presence in the room and Child Life Specialists in the room if desired), or the standard of care plus VR. Individuals assigned to the VR arm will be fitted with a Samsung head-tracking system, and will play an AppliedVR game prior to and during catheterization. Standardized questionnaires will be administered to patients and caregivers before and after the procedure to measure pain and anxiety. Satisfaction questionnaires will be administered post-procedure.

Significance: VR is a non-invasive intervention that, if effective, could become part of a standard protocol to reduce pain and anxiety among children undergoing VCUGs. As there is a dearth of knowledge regarding non-pharmacologic interventions for children receiving VCUGs, this study will provide a foundation to inform future research on VR use among pediatric urology patients.

See 'References' for Brief Summary References

ELIGIBILITY:
Inclusion criteria for children:

* Children who are 5-21 years old
* Children who are English or Spanish speaking.
* Children undergoing a VCUG at CHLA.
* Only children who are in the normal range of development will be recruited for this study. This will be assessed by report from the parents. The rationale for excluding patients with developmental delay is that due to their cognitive impairments, such children react to the stressors of medical procedures differently than do children without such developmental delay. It is unclear how such children would use the interventions included in this study, and it is likely that their responses on baseline and outcome measures will differ from children of normal developmental parameters.

Inclusion criteria for caregivers (no age limits):

* Have a child who is undergoing a VCUG at CHLA.
* Caregiver is present during the child's VCUG.
* Caregiver is English or Spanish speaking.
* Caregiver is 18 years old or older.

Inclusion criteria for healthcare providers (no age limits):

* Provider is 18 years old or older
* Provider is a CHLA employee.
* Provider may participate if he/she witnessed and/or administered the medical procedure.

Exclusion Criteria:

* Child is currently taking pain medication or anxiolytic medication, including midazolam
* Child has a psychiatric disorder (i.e. anxiety, psychotic, thought disorder), organic brain syndrome, intellectual disability, Autism Spectrum Disorder, or other known cognitive/neurological disorder
* Child has visual, auditory, or tactile deficit that would interfere with the ability to complete the experimental tasks
* Child has a history of seizure disorder
* Child is currently sick with flu-like symptoms or experiencing a headache or earache
* Child has known or suspected motion sickness
* Child catheterizes regularly or has an insensate urethra
* Languages other than English and Spanish will be excluded given that the proposed measures have not been standardized for use in other languages.

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 410 (Estimated)
Dates: Start 2020-02-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Pain during VCUG - Pain Visual Analog Scale | Will be administered to participants approximately 20 minutes before the start of the VCUG, and within 15 minutes following the end of the VCUG.
  Participant levels of pain will be assessed using the Pain Visual Analog Scale (min. score = 0; max. score = 100. Higher score = higher pain)

SECONDARY OUTCOMES:
Change in Pain during VCUG - Faces Pain Scale-Revised | Will be administered to participants approximately 20 minutes before the start of the VCUG, and within 15 minutes following the end of the VCUG.
  Participant levels of pain will be assessed using the Faces Pain Scale-Revised (min. score = 0; max. score = 10. Higher score = higher pain)
Change in Pain during VCUG - Colored Analog Scale | Will be administered to participants approximately 20 minutes before the start of the VCUG, and within 15 minutes following the end of the VCUG.
  Participant levels of pain will be assessed using the Colored Analog Scale (min. score = 0; max. score = 10. Higher score = higher pain)
Change in Anxiety during VCUG - Procedural Anxiety Visual Analog Scale | Will be administered to participants approximately 20 minutes before the start of the VCUG, and within 15 minutes following the end of the VCUG.
  Participant levels of anxiety will be assessed using the Procedural Anxiety Visual Analog Scale (min. score = 0; max. score = 10. Higher score = higher anxiety)
Change in Anxiety during VCUG - Facial Affective Scale | Will be administered to participants approximately 20 minutes before the start of the VCUG, and within 15 minutes following the end of the VCUG.
  Participant levels of anxiety will be assessed using the Facial Affective Scale (min. score = 0; max. score = 1. Higher score = higher anxiety)
Baseline Anxiety before VCUG - Anxiety Sensitivity Index | Will be administered to participants approximately 20 minutes before the start of the VCUG.
  Participant baseline anxiety will be assessed using the Anxiety Sensitivity Index, a 16-item questionnaire (min. score = 0; max. score = 64. Higher score = higher anxiety sensitivity; i.e. higher dispositional tendency to fear the somatic and cognitive symptoms of anxiety due to a belief that these symptoms may be dangerous or harmful).
Satisfaction with VR | Questionnaires will be administered to participants within 15 minutes following the end of the VCUG.
  Participant satisfaction with VR assessed using a 10-item satisfaction survey (min. score = 0; max. score = 50. Higher score = higher satisfaction).

CONTACTS AND LOCATIONS:
Overall Officials: Andy M Chang, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alexander M. Managing patient stress in pediatric radiology. Radiol Technol. 2012 Jul-Aug;83(6):549-60. PMID 22763832
- [Background] Guideline for Monitoring and Management of Pediatric Patients Before, During, and After Sedation for Diagnostic and Therapeutic Procedures: Update 2016. Pediatr Dent. 2016 Oct;38(6):216-245. PMID 27931463
- [Background] Glazer JD, Benrubi GI, Nuss RC. Positive results of endocervical curettage as an indication for conization of the cervix. South Med J. 1987 Feb;80(2):185-6. doi: 10.1097/00007611-198702000-00011. PMID 3810213
- [Background] Stashinko EE, Goldberger J. Test or trauma? The voiding cystourethrogram experience of young children. Issues Compr Pediatr Nurs. 1998 Apr-Jun;21(2):85-96. doi: 10.1080/014608698265519. PMID 10196917